CLINICAL TRIAL: NCT03218657
Title: A Prospective, Randomized, Controlled Clinical Study of Non Transfusion Dependent Non Severe Aplastic Anemia Treated With Cyclosporine, Androgen and Levamisole Hydrochloride
Brief Title: Clinical Study of Non Severe Aplastic Anemia Treated With Cyclosporine, Androgen and Levamisole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengyun Lin (Other)
Responsible Party: Sponsor-Investigator, Shengyun Lin, Chief, Zhejiang Provincial Hospital of TCM
Organization: Zhejiang Provincial Hospital of TCM (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA-LSA/SA
Record Dates: First submitted 2017-06-16; First posted 2017-07-14 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia; levamisole hydrochloride; clinical study
MeSH Terms: conditions — Anemia, Aplastic | interventions — Levamisole; Androgens; Cyclosporins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): the patients treated with levamisole hydrochloride 150mg qod +androgens 80mg qd+cyclosporins 3-5mg/kg*d at least for one year
  Interventions: Drug: levamisole hydrochloride; Drug: Androgens; Drug: Cyclosporins
- control group (Other): the patients treated without levamisole hydrochloride，but androgens 80mg qd+cyclosporins 3-5mg/kg*d at least for one year
  Interventions: Drug: Androgens; Drug: Cyclosporins

INTERVENTIONS:
Drug: levamisole hydrochloride — levamisole hydrochloride take orally 150mg qod
  Other Names: levamisole
  Arms: experimental group
Drug: Androgens — Androgens take orally 80mg qd
Drug: Cyclosporins — Cyclosporines take orally 3-5mg/kg*d qd

SUMMARY:
The clinical symptoms of non transfusion dependent non severe aplastic anemia (NSAA) are often lighter than that of severe aplastic anemia. Clinical observation is often used and the treatment should be given according to the follow-up results of peripheral blood routine and the survival condition of the patients. In recent years, a number of studies at home or abroad have tended to intervene earlier. The risk of observation and waiting for disease progression is higher. Early immunosuppression should be considered. For the treatment of non transfusion dependent non severe aplastic anemia, the commonly used treatment regimen is androgen combined with CSA. But the investigators find that Levamisole hydrochloride (LMS) as a commonly used immunomodulatory drugs may be helpful to improving immune disorder symptoms in NSAA patients. Therefore,the investigators are conducting a prospective, randomized controlled study to compare the rate, side effects and long-term survival in non transfusion dependent patients with NSAA between the androgen+CSA group and the androgen+CSA+LMS group.

ELIGIBILITY:
Inclusion Criteria:

1. All the patients meet a NSAA diagnostic criteria, and agree the immunosuppressive therapy. Diagnoses reference to The diagnostic and therapeutic criteria for hematologic diseases（Zhang Zhinan 2007）, and The diagnosis and treatment of aplastic anemia（2016 UK guidelines）
2. 18-70years old, male or female
3. Liver and kidney function: the blood bilirubin is less than or equal to 2mg/dL (35 mol/L), AST/ALT in the upper limit of the normal value below 2 times, blood inosine is less than or equal to 177 umol/L.
4. Heart function is normal: EF>50%.
5. No serious lung infection.
6. All cases had no history of cancer and chemotherapy history, immunology therapy. The control group without hematologic diseases, lupus or other immune disfunctions, allergic disease, Fanconi anemia.
7. Consent signed by patients or their families.

Exclusion Criteria:

1. Congenital hematopoietic failure, Fanconi anemia, or combined with bone marrow hyperplasia, leukemia, multiple myeloma, giant cell anemia, paroxysmal nocturnal hemoglobin or other blood diseases.
2. The HBV DNA copy number is greater than 1000/ml or the serum hepatitis B virus is not clear.
3. Serum bilirubin > 2mg/dL (35 umol/L); ALT or AST > 2 times the normal value of the upper limit; alkaline phosphatase > 3 times the upper limit of the normal value; serum creatinine > 177 mol/L.
4. HIV positive.
5. Other serious diseases that may limit the patient to participate in the study (e.g., the progressive infection, incontrollable diabetes, severe cardiac insufficiency or angina pectoris, etc.)
6. Conditions are not suitable for immunosuppressive therapy.
7. Pregnant or lactating women.
8. Can not understand or follow the research program.
9. Patients under 16 years of age.
10. Patients with a history of cancer, chemotherapy, or radiation therapy, immune system diseases or allergic diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Routine blood test | up to 4 weeks
  hemoglobin；white blood cell；Platelet

SECONDARY OUTCOMES:
Bone marrow | 1 year
  The proliferation of cells in bone marrow
biochemical test | up to 4 weeks
  Alanine aminotransferase；Aspartate aminotransferase

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Province Traditional Chinese Medical Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided